CLINICAL TRIAL: NCT03780452
Title: Use of Dynamic Intramedullary Compression Nail for Tibiocalcaneal Arthrodesis
Brief Title: Compression Nail for Tibiocalcaneal Arthrodesis
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: MedShape, Inc (Industry)
Responsible Party: Principal Investigator, Ashish Shah, Primary Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300002689
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Subtalar Arthritis; Ankle Arthritis
Keywords: intramedullary nail; arthrodesis; subtalar; tibiotalar
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tibiotalocalcaneal arthrodesis with DynaNail: Tibiotalocalcaneal arthrodesis with a novel dynamic compression intramedullary nail
  Interventions: Device: novel dynamic compression intramedullary nail

INTERVENTIONS:
Device: novel dynamic compression intramedullary nail — Tibiotalocalcaneal (TTC) arthrodesis with a novel dynamic compression intramedullary nail. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a novel dynamic compression intramedullary nail for tibiotalocalcaneal (TTC) arthrodesis

DETAILED DESCRIPTION:
This proposal is a collaborative effort of MedShape Inc. It is a prospective investigation to assess the clinical outcomes of patients with a tibiotalocalcaneal arthrodesis with the Dynamic Compression Intramedullary Nail (DynaNail). We are planning to enroll 30 patients. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

Patients with end-stage tibiotalar (ankle) and talocalcaneal (subtalar) joint arthritis from any etiology will be asked to enroll in the study. After informed consent, the patients will be asked to complete the following patient reported outcomes questionnaires (standard of care for all patients in the Foot and Ankle section): 100mm VAS for pain, Short form-36 (SF-36), and the Foot and Ankle Ability Measure (FAAM). After informed consent, they will then be scheduled for surgery in a routine fashion. REDCap database will be used to allow on-line data entry.

The following surgical procedure steps and follow-ups are standard of care at the University of Alabama at Birmingham. The surgical procedure will involve both tibiotalar and talocalcaneal joint preparation through any approach (lateral, posterior, anterior with sinus tarsi). The use of supplemental bone graft is at the discretion of the treating surgeon but must be documented. The MedShape DynaNail will then be inserted according to the manufacturer's technique. The patient will be placed in a short leg splint and kept non-weight bearing. The patient will be discharged from the hospital when medically ready and follow-up in two weeks.

At two weeks, the patient will return to clinic for a standard of care visit and their splint will be removed. A non-weight bearing lateral radiograph of the hind foot will be taken to assess the amount of travel of the compressive element. This radiograph is not standard of care. The patient will be placed in a non-weight bearing cast. The patient will then be asked to return in two weeks (4 weeks post-operatively). This visit is not standard of care. At this time another non-weight bearing lateral radiograph will be taken to assess the amount of travel of the compressive element. The patient will be asked to return at 6 weeks, 3 months, 6 months, 12 months, and 24 months after surgery as is standard of care for this surgery. At each of these time-points, the same patient specific outcome questionnaires will be administered. For any non- standard of care radiographs patients will be asked to take a urine pregnancy test prior to any radiographs being taken.

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon, his clinical fellow, or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the only exclusion criteria will be patients who are not healthy enough to undergo surgery. Patients of all racial, religious, and cultural backgrounds will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Ankle and Subtalar arthritis
* Failed non-operative management

Exclusion Criteria:

* Patients who do not meet the minimum age of 18 years.
* patients who are not eligible to undergo surgery

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon, his clinical fellow, or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the only exclusion criteria will be patients who are not healthy enough to undergo surgery. Patients of all racial, religious, and cultural backgrounds will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ashish shah, md, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited if they met the indications for tibiotalocalcaneal arthrodesis, were able to understand the requirements of the study, provide a written consent, and were willing to comply with the study protocol, and were over 18 years of age. Patients were recruited between 2020 and 2023 at an Orthopedic Clinic at a busy urban medical center.
Pre-assignment Details: Patients were screened for those scheduled to undergo a tibiotalocalcaneal arthrodesis at an ambulatory surgery center with one of the participating foot and ankle fellowship trained orthopaedic surgeons. Patients enrolled in the study had their surgery performed with a Dynamic compression Intramedullary Nail with the aim of improved function and pain. Follow-up occurred in clinic and via surveys pre-operatively, as well as, 2-weeks, 6-weeks, 12-weeks, 24-weeks, and 1 year post-operatively
Groups:
- Tibiotalocalcaneal Arthrodesis With DynaNail: Tibiotalocalcaneal arthrodesis with a novel dynamic compression intramedullary nail
  novel dynamic compression intramedullary nail: Tibiotalocalcaneal (TTC) arthrodesis with a novel dynamic compression intramedullary nail. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.
  Patients were screened for those scheduled to undergo a tibiotalocalcaneal arthrodesis at an ambulatory surgery center with one of the participating foot and ankle fellowship trained orthopaedic surgeons. Patients enrolled in the study had their surgery performed with a Dynamic compression Intramedullary Nail with the aim of improved function and pain. Follow-up occurred in clinic and via surveys pre-operatively, as well as, 2-weeks, 6-weeks, 12-weeks, 24-weeks, and 1-year post-operativel
Period: Overall Study
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Started | 13
Completed | 11
Not Completed | 2
Not completed — Screening failure | 2

BASELINE CHARACTERISTICS:
Population: Population is the same as listed in Participant Flow.
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  BMI < 30 | 3
  BMI > = 30 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment
Description: Visual Analog Scale (VAS). Patients will disclose their pain level using the Visual Analog Scale, which measures pain on a scale of 0 - 100, with 0 indicating no pain and 100 indicating severe pain.
Time Frame: 0 - 12 months postoperatively
Population: Patients having undergone tibiotalocalcaneal arthrodesis with completion of Visual Analog Scale surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Number analyzed (Participants) | 11
score on a scale
  Baseline | 52.73 (22.60)
  2 Weeks | 33.00 (30.35)
  6 Weeks | 17.00 (26.19)
  12 Weeks | 21.25 (26.19)
  24 Weeks | 20.00 (15.11)
  1 Year | 34.00 (25.77)

2. Primary Outcome: Functional Assessment
Description: Foot and Ankle Ability Measure (FAAM). The FAAM is made up of a 21-item activity of daily living (ADL) and and 8-item sports subscale, which are combined to form a single total score. The ADL subscale ranges from 0 to 84 and the sports from 0 to 32. The total score is a calculated by adding the two subscores together and then reporting as a percentage of the total possible score (116). The percent score range is from 0% to 100%. For interpretation of the results a score closure to 100% is considered greater function.
Time Frame: 0 - 12 months postoperatively
Population: Patients analyzed include those that underwent tibiotalocalcaneal arthrodesis with a Dynamic Compression Intramedullary Nail who completed their Foot and Ankle Ability Measure surveys.
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Number analyzed (Participants) | 11
percentage of total score
  Baseline | 48.18 (36.32)
  2 Weeks | 42.27 (60.95)
  6 Weeks | 14.55 (16.53)
  12 Weeks | 56.00 (50.79)
  24 Weeks | 77.85 (60.29)
  1 Year | 53.5 (3.5)

3. Primary Outcome: Change in Functional Assessment
Description: The Short Form 36 (SF-36) is a total of 36 questions covering 8 domains of health: (1) limitations in physical activities, (2) limitations in social activities, (3) limitations in usual role activities due to physical health problems, (4) bodily pain, (5) general mental health, (6) Limitations in usual role activities due to emotional problems, (7) Vitality, and (8) General health perceptions. The domain scores are added together for a total score. The total is a reported as a percentage from 0% to 100% with 50 serving as the normative value. Higher scores represent a greater level of functioning.
Time Frame: 0 - 12 months postoperatively
Population: Patients analyzed include those that underwent tibiotalocalcaneal arthrodesis with a Dynamic Compression Intramedullary Nail who completed their Short Form 36 surveys.
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Number analyzed (Participants) | 11
percentage of total score
  Baseline | 24.74 (12.78)
  2 Weeks | 23.82 (12.25)
  6 Weeks | 27.46 (15.00)
  12 Weeks | 37.64 (9.68)
  24 Weeks | 40.56 (12.64)
  1 Year | 39.64 (8.73)

4. Primary Outcome: Fusion, as Measured by Radiograph and CT Scan
Description: radiographs taken Pre-operatively, 2 weeks, 4 weeks, 6 weeks, 3 Months, 6 Months, 12 Months and 24 Months. A CT scan will be done at 6 months.
Time Frame: 0 - 12 months postoperative
Population: Patients analyzed include those that underwent tibiotalocalcaneal arthrodesis with a Dynamic Compression Intramedullary Nail with post-operative imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
Number analyzed (Participants) | 8
Participants
  Union | 7
  Nonunion | 1
  Malunion | 0

ADVERSE EVENTS:
Time Frame: 0-12 months post-operative
Arm/Group | Tibiotalocalcaneal Arthrodesis With DynaNail
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tibiotalocalcaneal Arthrodesis With DynaNail (N=11)
Implant Failure (Product Issues) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03780452/Prot_SAP_000.pdf